CLINICAL TRIAL: NCT06482996
Title: the Impact of General Anesthesia on Blood Pressure and Intraocular Pressure in Geriatric Patients Undergoing Cataract Surgery
Brief Title: General Anesthesia on Blood Pressure and Intraocular Pressure in Geriatric Patients Undergoing Cataract Surgery
Status: Recruiting | Type: Observational
Sponsor: Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Zeliha Alicikus, head of Anesthesia and reanimation, Umraniye Education and Research Hospital
Other Study IDs: UERH-AR-ZT-08
Record Dates: First submitted 2024-05-06; First posted 2024-07-01 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Cataract
Keywords: Cataract surgery; Frailty
MeSH Terms: conditions — Cataract; Frailty | interventions — Intraocular Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group A: Frail scale:Non frail
  Interventions: Other: Intraocular pressure (IOP) was measured
- group B: Frail scale: Pre frail/frail
  Interventions: Other: Intraocular pressure (IOP) was measured

INTERVENTIONS:
Other: Intraocular pressure (IOP) was measured — The Frail Scale was used to assess the frailty of the patients.Intraocular pressure (IOP) was measured before anesthesia, 5 minutes after induction of anesthesia and 1 hour postoperatively. IOP was measured using a Tono-pen tonometer (AccuPen). The normal range of IOP is 11-21 mmHg (mean 16 mmHg) and values above 24 mmHg are pathologic.

SUMMARY:
The primary aim of the study is to investigate the correlation between preoperative hemodynamics and frailty scores in patients undergoing cataract surgery under general anesthesia. The secondary objective is to explore the relationship between preoperative and postoperative intraocular pressure changes and frailty scores.

DETAILED DESCRIPTION:
Cataract stands as a significant cause of vision impairment worldwide, notably prevalent among the elderly. This study aims to explore the changes in intraocular pressure (IOP) and blood pressure under general anesthesia during cataract surgery in frail geriatric patients. The research emphasizes the critical role of frailty assessment in determining surgical risks among elderly surgical patients. It focuses on the hypothesis that frail individuals undergoing cataract surgery under general anesthesia might experience more pronounced effects on IOP and blood pressure during the surgical procedure compared to prefrail counterparts. This study emerges as a crucial step in understanding the impact of preoperative frailty assessment on surgical planning and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 65-85 age
* ASA I-III
* cataract surgery with genel anesthesia

Exclusion Criteria:

* cerebrovascular disease,
* mental retardation and psychiatric illness,
* pulmonary infection, history of advanced COPD or respiratory failure,
* EF less than 40%, presence of cardiovascular disease,
* bleeding diathesis,
* renal and hepatic insufficiency,
* presence of diabetes mellitus, diuretic/mannitol users,
* substance abuse
* BMI >30

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: This prospective randomized controlled double-blind study included a total of 80 ASA I-III patients aged 65-85 years undergoing cataract surgery under general anesthesia. Randomization Patients were randomly divided into two groups with frailty score as non-frail (40 patients) and pre-frail/frail (40 patients) by closed envelope method.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-02-27 (Estimated)

PRIMARY OUTCOMES:
intraocular pressure during genel anesthesia | through study completion, an average of 1 day
  intraocular pressure (mmHg)

SECONDARY OUTCOMES:
hemodynamic data | through study completion, an average of 1 day
  mean arterial pressure (mmHg)

CONTACTS AND LOCATIONS:
Locations (1):
- Umraniye Education and Research hospital, Istanbul, Turkey (Türkiye)